CLINICAL TRIAL: NCT01487733
Title: Analysis of HPV and Other Biomarkers in Specimens From ECOG Studies in Recurrent or Metastatic Head and Neck Cancer (E1395 and E3301)
Brief Title: Biomarkers in Tissue Samples From Patients With Recurrent or Metastatic Head and Neck Cancer Treated on ECOG-E1395 and ECOG-E3301
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000717143; ECOG-E4L10T1
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IVA squamous cell carcinoma of the larynx; stage IVA squamous cell carcinoma of the lip and oral cavity; stage IVA squamous cell carcinoma of the oropharynx; stage IVA squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVB squamous cell carcinoma of the larynx; stage IVB squamous cell carcinoma of the lip and oral cavity; stage IVB squamous cell carcinoma of the oropharynx; stage IVB squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVC squamous cell carcinoma of the larynx; stage IVC squamous cell carcinoma of the lip and oral cavity; stage IVC squamous cell carcinoma of the oropharynx; stage IVC squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IVA salivary gland cancer; stage IVB salivary gland cancer; stage IVC salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Gene Expression Profiling; In Situ Hybridization; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: in situ hybridization
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with recurrent or metastatic head and neck cancer treated on ECOG-E1395 and ECOG-E3301.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the association between biomarkers (HPV tumor status and ERCC1 expression) and clinical outcomes in a population of patients with recurrent or metastatic head and neck cancer.
* To develop the ability to select patients likely to respond to therapy and to avoid treatment with ineffective therapies, especially since these therapies have substantial toxicity.
* To estimate response and survival rates of HPV-negative and -positive patients in each study. (exploratory)

OUTLINE: Tumor HPV status is determined by in situ hybridization (ISH) and all samples also undergo immunostaining for p16. ERCC1 expression is evaluated with AQUA, a quantitative IHC analysis.

Samples are classified into two categories based on their biomarker status: HPV tumor status (negative versus positive), and ERCC1 expression level (low versus high).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tissue specimens from patients with recurrent or metastatic head and neck cancer treated on ECOG-E1395 and ECOG-E3301

  * Stage III, IV, or recurrent disease
  * Squamous cell disease
  * Any of the following diagnoses:

    * Lip and oral cavity
    * Oropharynx
    * Hypopharynx
    * Larynx
    * Paranasal sinus and nasal cavity
    * Squamous neck cancer
    * Salivary gland

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients who participated in E1395 or E3301 and provided samples for research.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2011-12-22 (Actual); Primary Completion 2012-01-22 (Actual); Study Completion 2012-01-22 (Actual)

PRIMARY OUTCOMES:
Treatment response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio

REFERENCES:
- [Derived] Argiris A, Li S, Ghebremichael M, Egloff AM, Wang L, Forastiere AA, Burtness B, Mehra R. Prognostic significance of human papillomavirus in recurrent or metastatic head and neck cancer: an analysis of Eastern Cooperative Oncology Group trials. Ann Oncol. 2014 Jul;25(7):1410-1416. doi: 10.1093/annonc/mdu167. Epub 2014 May 5. PMID 24799460